CLINICAL TRIAL: NCT04182334
Title: Decreasing Delirium Through Music in Critically Ill Older Adults
Acronym: DDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1906664366; 5R01AG067631-03 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care Unit Delirium; Pain; Anxiety; Intensive Care Acquired Cognitive Impairment
Keywords: Delirium; Music; Pain; Anxiety; Cognition
MeSH Terms: conditions — Pain; Anxiety Disorders; Delirium

STUDY DESIGN:
Intervention Model Description: Slow Tempo Music vs Attention Control
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the unblinded study coordinator is aware of randomization. Outcomes assessors are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow Tempo Music (Experimental): Slow-tempo 60-80 beats per minute relaxing music. The intervention includes two one-hour music listening sessions, once in the morning and once in the evening for up to seven days, delivered through noise-canceling headphones and iPad.
  Interventions: Other: Slow Tempo Music
- Attention Control (Sham Comparator): One-hour sessions consisting of a silence track twice daily delivered through noise-cancelling headphones for up to 7 days.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Slow Tempo Music — For up to seven days, enrolled subjects will receive one-hour slow tempo music listening sessions twice daily through noise-cancelling headphones.
  Arms: Slow Tempo Music
Other: Attention Control — Subjects will receive a noise cancellation headphone-applied condition identical to the music intervention experimental treatment in twice daily one hour-sessions for up to seven days.
  Arms: Attention Control

SUMMARY:
Critically ill older adults admitted to the intensive care unit (ICU) are at a higher risk to develop delirium, which predisposes them to longer lengths of ICU and hospital stay, increased in-patient mortality, and higher risk of new acquired cognitive impairment and dementia. Music listening is a non-pharmacological intervention that holds potential to decrease ICU delirium. The investigators propose a randomized controlled trial to evaluate the efficacy of a seven-day slow-tempo music intervention on the primary outcome of delirium/coma free days among mechanically ventilated, critically ill older adults.

DETAILED DESCRIPTION:
One million adults in the United States receive mechanical ventilation for acute respiratory failure in the intensive care units (ICUs) annually and up to 80% of them develop delirium during their ICU stay. Presence of delirium predisposes older adults to immediate in-hospital complications including a longer length of ICU and hospital stay, increased risk of in-patient mortality and elevated costs of care. In addition, ICU delirium is associated with long-term post-discharge complications such as development of cognitive impairment and dementia.

Recent research studies exploring pharmacological strategies to manage ICU delirium have not demonstrated efficacy; a limitation also acknowledged in the Society of Critical Care Medicine 2018 Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption guidelines. Music listening is a non-pharmacological intervention that has shown to decrease over-sedation, anxiety and stress in critically ill patients, factors that could predispose to ICU delirium. Our team is now proposing to conduct a large randomized clinical trial called "Decreasing Delirium through Music (DDM) in Critically Ill Older Adults to evaluate the efficacy of a seven-day slow-tempo music intervention on the primary outcome of delirium/coma free days among mechanically-ventilated older adults admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years or older.
2. English speaking.
3. Admitted to the intensive care unit (medical or surgical).
4. Expected mechanical ventilator support for ≥48 hours.
5. Consentable through a legally authorized representative.
6. Have access to a telephone.

Exclusion Criteria:

1. History of dementing illnesses and other neurodegenerative diseases such as Alzheimer's disease or vascular dementia.
2. Psychiatric illness which is not well controlled.
3. Alcohol withdrawal symptoms/concern for withdrawal.
4. Suspected or confirmed drug intoxication/overdose
5. Traumatic brain injury, ischemic or hemorrhagic cerebrovascular accident, or undergoing neurosurgery.
6. Uncorrected hearing or vision impairment including legal blindness.
7. Incarcerated at the time of study enrollment.
8. Enrolled in another clinical trial which does not permit co-enrollment.
9. Any medical condition precluding safe use of headphones such as: skin breakdown, burns, facial or skull fractures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babar Khan, MD, MS, Principal Investigator — Indiana University; Linda Chlan, PhD, RN, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - IU Health West Hospital, Avon, Indiana
  - Eskenazi Hospital, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan BA, Khan SH, Perkins AJ, Heiderscheit A, Unverzagt FW, Wang S, Downs JH 3rd, Gao S, Chlan LL. Slow-Tempo Music and Delirium/Coma-Free Days Among Older Adults Undergoing Mechanical Ventilation: A Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 1;185(12):1442-1453. doi: 10.1001/jamainternmed.2025.5263. PMID 41082215
- [Derived] Seyffert S, Moiz S, Coghlan M, Balozian P, Nasser J, Rached EA, Jamil Y, Naqvi K, Rawlings L, Perkins AJ, Gao S, Hunter JD 3rd, Khan S, Heiderscheit A, Chlan LL, Khan B. Decreasing delirium through music listening (DDM) in critically ill, mechanically ventilated older adults in the intensive care unit: a two-arm, parallel-group, randomized clinical trial. Trials. 2022 Jul 19;23(1):576. doi: 10.1186/s13063-022-06448-w. PMID 35854358

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol subjects were considered to be enrolled in the study at the time of completion of the informed consent process. 160 subjects were enrolled. 159 subjects were randomized to one of the two study groups.
Period: Overall Study
Arm/Group | Slow Tempo Music | Attention Control
Started | 79 | 80
Completed | 59 | 55
Not Completed | 20 | 25

BASELINE CHARACTERISTICS:
Population: 160 subjects were enrolled, 159 subjects were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Slow Tempo Music | Attention Control | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.1) | 68.2 (9.3) | 67.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 45 | 42 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 15 | 30
  White | 59 | 63 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Days Free of Delirium and Coma
Description: Days free of delirium and coma will be the primary outcome for the trial. Days free of delirium and coma are the number of days after randomization patient is alive free of delirium and not in coma during the seven-day study intervention phase.
Time Frame: Seven day study intervention phase
Measure: Median (Full Range); unit: Delirium/coma-free days by day 7
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 79 | 80
Delirium/coma-free days by day 7 | 2.5 [0 to 5] | 3 [0 to 5]
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.775, Mixed Models Analysis

2. Secondary Outcome: Delirium Severity
Description: Delirium severity was assessed twice daily by trained research assistants by the CAM-ICU-7, a seven point rating scale (0-7) where higher scores reflect higher delirium severity (worse outcomes). The CAM-ICU-7 score are categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium. For the twice daily assessments, the mean of the two assessments was used.
Time Frame: Subjects will be followed up to 28 days post randomization. The first 7 days were used for analysis per the protocol statistical plan.
Population: maximum number of participants analyzed during day 1 through day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 68 | 67
score on a scale
  Day 1 | 5.43 (2.35) | 5.79 (2.16)
  Day 2: number analyzed (Participants) | 67 | 67
  Day 2 | 4.77 (2.35) | 5.51 (2.18)
  Day 3: number analyzed (Participants) | 62 | 65
  Day 3 | 4.10 (2.55) | 4.45 (2.61)
  Day 4: number analyzed (Participants) | 56 | 55
  Day 4 | 3.54 (2.75) | 3.95 (2.72)
  Day 5: number analyzed (Participants) | 47 | 52
  Day 5 | 2.78 (2.70) | 3.27 (2.83)
  Day 6: number analyzed (Participants) | 45 | 44
  Day 6 | 2.73 (2.73) | 3.49 (2.94)
  Day 7: number analyzed (Participants) | 43 | 42
  Day 7 | 2.72 (2.80) | 2.56 (2.72)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.995, Mixed Models Analysis

3. Secondary Outcome: Pain Intensity
Description: Pain will be assessed by trained research assistants utilizing the Critical Care Pain Observation Tool (CPOT), a valid and reliable instrument in critically ill patients with and without delirium.. Scale range 0-8, higher score indicates worse pain. For the 4 times daily assessments, the mean of the 2 post intervention assessments was used.
Time Frame: 4 times daily, before and after each intervention for up to 7 days while in the ICU and then twice daily up to 28 days post randomization. The first 7 days were used for analysis per the protocol statistical plan.
Population: maximum number of participants analyzed during day 1 through day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 67 | 66
score on a scale
  Day 1 | 0.42 (0.94) | 0.30 (0.72)
  Day 2: number analyzed (Participants) | 67 | 62
  Day 2 | 0.34 (0.85) | 0.34 (0.83)
  Day 3: number analyzed (Participants) | 52 | 50
  Day 3 | 0.32 (0.82) | 0.21 (0.47)
  Day 4: number analyzed (Participants) | 44 | 43
  Day 4 | 0.51 (0.87) | 0.31 (0.65)
  Day 5: number analyzed (Participants) | 31 | 32
  Day 5 | 0.44 (0.91) | 0.31 (0.64)
  Day 6: number analyzed (Participants) | 24 | 26
  Day 6 | 0.17 (0.48) | 0.25 (0.47)
  Day 7: number analyzed (Participants) | 22 | 19
  Day 7 | 0.20 (0.55) | 0.61 (1.29)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.674, Mixed Models Analysis

4. Secondary Outcome: Anxiety
Description: Anxiety intensity defined as a heightened state of apprehension, agitation, and arousal, will be measured four times daily before and after assigned intervention using a 100-mm Visual Analog Scale-Anxiety (VAS-A). Scale range 0-100, higher score indicates worse anxiety. For the 4 times daily assessments, the mean of the 2 post intervention assessments was used.
Time Frame: as for outcome 3
Population: maximum number of participants analyzed during day 1 through day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 25 | 19
score on a scale
  Day 1: number analyzed (Participants) | 16 | 8
  Day 1 | 40.56 (34.41) | 43.13 (33.77)
  Day 2: number analyzed (Participants) | 25 | 17
  Day 2 | 38.40 (33.49) | 38.82 (34.81)
  Day 3 | 39.38 (37.45) | 35.39 (38.28)
  Day 4: number analyzed (Participants) | 21 | 15
  Day 4 | 37.86 (36.36) | 39.50 (33.31)
  Day 5: number analyzed (Participants) | 16 | 13
  Day 5 | 25.72 (30.23) | 53.50 (38.97)
  Day 6: number analyzed (Participants) | 11 | 10
  Day 6 | 34.36 (35.40) | 37.80 (44.57)
  Day 7: number analyzed (Participants) | 8 | 6
  Day 7 | 43.63 (24.67) | 28.83 (38.40)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.326, Mixed Models Analysis

5. Secondary Outcome: Cognition
Description: Cognition will be measured by objective tests of memory, attention, information processing speed and executive cognitive function. The Auditory Verbal Learning Test [AVLT] will be administered using a phone-based format. During test administration there are 5 learning trials. After a 30-minute delay, the participants are asked to recall as many words as possible. The sum of learning trials are presented as scores ranging from 0-75, and for the 30-minute delay test scores range from 0-15. A lower score indicates a worse outcome.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 13 | 17
score on a scale
  AVTL Total Learning | 32.23 (13.14) | 35.76 (12.10)
  AVTL Delayed Recall | 5.3 (3.6) | 5.9 (3.4)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.463, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Cognition
Description: Cognition will be measured by objective tests of memory, attention, information processing speed and executive cognitive function. The Wechsler Adult Intelligence Scale- III Digit Span test will be administered using a phone-based format. Score range 0-30, a lower score indicates a worse outcome.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 13 | 17
score on a scale | 15.85 (6.08) | 13.88 (4.48)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.449, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Cognition
Description: Cognition will be measured by objective tests of memory, attention, information processing speed and executive cognitive function. The Symbol Digit Modalities Test will be administered using a phone-based format. Score range 0-110, a lower score indicates a worse outcome.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 10 | 15
score on a scale | 35.10 (21.08) | 30.13 (12.44)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.505, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Cognition
Description: Cognition will be measured by objective tests of memory, attention, information processing speed and executive cognitive function. The Multilingual Aphasia Examination Controlled Oral Word Association test will be administered using a phone-based format. Score range 0-no max score, a lower score indicates a worse outcome.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 13 | 15
score on a scale | 32.31 (14.46) | 34.13 (10.22)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.612, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Depression
Description: We will use the Patient Health Questionnaire-9 (PHQ-9) to determine the impact of the music intervention on ICU survivor's mood. Scale range 0-27, higher score indicates worse depression.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 13 | 16
score on a scale | 3.38 (3.62) | 7.50 (6.39)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.058, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Anxiety
Description: We will use the Generalized Anxiety Disorder Scale (GAD-7) to determine the impact of the music intervention on ICU survivor's anxiety. Scale range 0-21, higher score indicates worse anxiety.
Time Frame: 3 months post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Slow Tempo Music | Attention Control
Number analyzed (Participants) | 13 | 16
score on a scale | 2.46 (2.85) | 5.94 (6.49)
Statistical Analysis 1: Comparison: Slow Tempo Music vs Attention Control; Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from the time of informed consent process completion until the end of study participation. This was approximately 1 year if the study was completed.
Arm/Group | Slow Tempo Music | Attention Control
All-Cause Mortality (participants affected / at risk) | 10/79 | 10/80
Serious Adverse Events (participants affected / at risk) | 1/79 | 0/80
Other Adverse Events (participants affected / at risk) | 2/79 | 2/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Tempo Music (N=79) | Attention Control (N=80)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Tempo Music (N=79) | Attention Control (N=80)
Hallucination (Nervous system disorders) | 1 (1) | 0 (0)
Ear/ earlobe skin breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04182334/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04182334/ICF_001.pdf